CLINICAL TRIAL: NCT06553313
Title: Analysis of Protein Expression in Serum of Subjects With Knee Arthritis Control Group and Evaluation by Meridian and Pulse Wave Energy
Brief Title: Analysis of Protein Expression in Serum of KOA Subjects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CMUH113-REC3-115
Record Dates: First submitted 2024-08-04; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Enzyme-Linked Immunosorbent Assay

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the control group of knee arthritis (Other): Monitoring the stability of protein expression, pulse wave and meridian energy in the serum of the KOA control group (participants without knee pain).
  Interventions: Device: Micro-Western Array

INTERVENTIONS:
Device: Micro-Western Array — The subjects first took the energy measurement of the pulse sphygmograph and Ryodoraku, rested for 20 minutes, and then repeated the measurements again. In order to comply with the acupuncture treatment course was 5 weeks in the previous study, we have two blood draw point. Each subject's blood was drawn for the first time, and then for the second time in 5 weeks later. Each subject drew 10ml of blood each time. The blood samples are analyzed by Micro-Western Array (MWA) and Enzyme-linked immunosorbent assay (ELISA) to obtain the serum protein content value of healthy individuals.
  Other Names: Enzyme-linked immunosorbent assay; pulse sphygmograph; Ryodoraku

SUMMARY:
In the previous study "Using omics technology to explore the mechanism of acupuncture treatment of different acupoints of knee osteoarthritis: a randomized controlled trial (CMUH109-REC3-113)", we found that acupuncture for knee osteoarthritis(KOA) significantly reduces inflammation, apoptosis, and metabolism-related serum protein profiles. However, due to the lack of serum protein data from the control group, it is impossible to establish standard values for comparison. To analyze the protein expression in the serum of KOA control group subjects, we also measured the spectral energy values of the radial artery pulse wave obtained from the pulse sphygmograph and the meridian energy values obtained from Ryodoraku. The results obtained can be compared with previous studies, thus this experiment was designed.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 50 years old without knee pain

Exclusion Criteria:

1. Clinical diagnosis of knee osteoarthritis
2. Taking anti-inflammatory and analgesic drugs in the past month
3. Taking blood-lipid-lowering drugs or health foods in the past month
4. Received any acupuncture treatment in the past 3 weeks

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-04 (Actual); Primary Completion 2025-07-23 (Estimated); Study Completion 2025-07-23 (Estimated)

PRIMARY OUTCOMES:
Micro-Western Array and Enzyme-linked immunosorbent assay | the first and the fifth weeks
  Obtaining the serum protein content value

SECONDARY OUTCOMES:
pulse sphygmograph and Ryodoraku | the first and the fifth weeks
  the energy measurement of pulse and meridians

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Zhen Yu, Principal Investigator — China Medical University, China
Locations (1):
- China Medical University, Taichung, Taiwan